CLINICAL TRIAL: NCT00888420
Title: The Application of Performance Improvement Principles to the Patient Throughput Process in an Adult Outpatient Pain Treatment Clinic
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Thomas R. Vetter, MD, MPH, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: X080201003
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Pain
Keywords: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Medical Management: Patient satisfaction under current operational conditions
- Interventional Management: Patient satisfaction under the PSDA (Plan, do, study, act) performance improvement measures
  Interventions: Other: Performance Improvement Measures

INTERVENTIONS:
Other: Performance Improvement Measures — PDSA (Plan, Do, Study, Act) performance improvement measures
  Groups: Interventional Management

SUMMARY:
This study is undertaken to assess and improve the existing patient flow, or so-called throughput process, in an adult outpatient pain treatment clinic.

ELIGIBILITY:
Inclusion Criteria:

* 19-100 years of age.
* patient presenting to the UAB Highlands Pain Treatment Clinic for initial evaluation and treatment or subsequent follow-up evaluation and treatment.

Exclusion Criteria:

* <19 or >100 years of age
* a current prisoner

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient pain clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 1221 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
the total time patients spend to receive chronic pain treatment | prospective

SECONDARY OUTCOMES:
The total time health care providers must devote to delivering chronic pain treatment | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Vetter, MD, MPH, Principal Investigator — UAB Department of Anesthesiology
Locations (1):
- UAB Highlands Pain Treatment Clinic, Birmingham, Alabama, United States